CLINICAL TRIAL: NCT01329692
Title: Early Intervention in Patients With Predicted Poor Long-term Outcome Following Laparoscopic Roux-en-Y Gastric Bypass: a Prospective Randomized Study
Brief Title: Early Intervention for Morbidly Obese Patients After Roux-en-Y Gastric Bypass (RYGB) Surgery
Acronym: Back on Track
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI has left Duke-the primary study site and the sponsor retreat the support
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: Pro00025927
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Weight Loss; Obesity
Keywords: RYGB; Intervention; follow-up; standard-of-care; Back on Track program; poor weight loss; morbidly obese
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): This is a seven-week group education, counseling, nutrition, exercise, and journaling program of the Duke Metabolic and Weight Loss Surgery Center designed to help postoperative bariatric surgery patients who are failing to progressively lose weight resume an expected pattern of weight loss and improved overall outcome.
  Weeks 1 and 2 consist primarily of a review of current dietary habits. Weeks 3, 4, & 5 introduces counseling, with specific emphasis on emotional aspects of eating and behavioral modification strategies. Week 6 focuses on the metabolic impact of exercise, and includes an exercise session with a personal trainer. Week 7 incorporates a question and answer session with a sharing of discoveries, as well as an option for additional individual follow-up as needed.
  Interventions: Behavioral: Lifestyle counseling
- RYGB regular post-op care (No Intervention): Regular care and follow-up after RYGB surgery

INTERVENTIONS:
Behavioral: Lifestyle counseling — Weeks 1 and 2 consist primarily of a review of current dietary habits with initiation of a food journal; a basic review of macronutrients and metabolism; and the beginning of a weekly exercise regimen. Weeks 3, 4, & 5 introduces counseling, with specific emphasis on emotional aspects of eating and behavioral modification strategies. Week 6 focuses on the metabolic impact of exercise, and includes an exercise session with a personal trainer. Week 7 incorporates a question and answer session with a sharing of discoveries, as well as an option for additional individual follow-up as needed. During this period, patients will also be given access to an interactive web-based tool providing additional emphasis on the aforementioned components and clinician follow-up.
  Arms: Lifestyle counseling

SUMMARY:
Purpose and objective: To identify in the early post-operative period following laparoscopic Roux-en-Y gastric bypass patients likely to fail to progressively lose weight in expected fashion, and to institute intervention and assess for its efficacy.

Study activities and population group: Patients identified to have "poor weight loss" (≤ 11% of excess weight loss) at 1 month will be randomized into a control versus study group. Intervention for subjects randomized to the IV arm will be by enrollment in the Back on Track program. This is a seven-week group education, counseling, nutrition, exercise, and journaling program of the Duke Weight Loss Surgery Center designed to help postoperative bariatric surgery patients who are failing to progressively lose weight resume an expected pattern of weight loss and improved overall outcome.

Data analysis and risk/safety: Data will be collected and analyzed by the identified investigators. The goal of data analysis is to uncover any difference in the EWL of subjects who underwent intervention for falling in the lowest EWL quartile when compared with those who did not undergo intervention, and determine the statistical significance of any such difference. There are no physical risks associated with this study. There is, however, the potential risk of loss of confidentiality. Every effort will be made to keep your information confidential.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Patient is scheduled and consented for laparoscopic Roux-en-Y gastric bypass as part of their routine medical care

Exclusion Criteria:

* Younger than Age 18 years
* Patient is disabled and unable to participate in an exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
First quartile excess weight loss(0-11% EWL)at one month predicted first quartile EWL at 12-month and 36-month follow-up. | 1-7 week intervention, 3,6, and 12 months follow-up
  Weeks 1 and 2 consist primarily of a review of current dietary habits. Weeks 3, 4, & 5 introduces counseling, with specific emphasis on emotional aspects of eating and behavioral modification strategies. Week 6 focuses on the metabolic impact of exercise, and includes an exercise session with a personal trainer. Week 7 incorporates a question and answer session with a sharing of discoveries, as well as an option for additional individual follow-up as needed.

CONTACTS AND LOCATIONS:
Locations (1):
- Durham Regional Hospital, Durham, North Carolina, United States